CLINICAL TRIAL: NCT04239508
Title: Swiss Neonatal Network & Follow-up Group
Acronym: SwissNeoNet
Status: Recruiting | Type: Observational
Sponsor: Swiss Neonatal Network (Network)
Collaborators: Department of Neonatology, Children's Clinic, Cantonal Hospital Aarau, Switzerland (Unknown); Department of Neuropaediatrics, Children's Clinic, Cantonal Hospital Aarau, Switzerland (Unknown); Department of Neonatology, University of Basel Children's Hospital (UKBB), Switzerland (Unknown); Department of Neuropaediatrics and Developmental Medicine, University of Basel Children's Hospital (UKBB), Switzerland (Unknown); Department of Pediatrics, San Giovanni Hospital Bellinzona, Switzerland (Unknown); Department of Neonatology, University Hospital Berne, Switzerland (Unknown); Department of Neuropaediatrics, University Hospital Berne, Switzerland (Unknown); Development and Pediatric Neurorehabilitation Center, Biel, Switzerland (Unknown); Department of Neonatology, Children's Hospital Chur, Switzerland (Unknown); Department of Neuropaediatrics, Children's Hospital Chur, Switzerland (Unknown); Department of Neuropediatrics, Cantonal Hospital Fribourg, Switzerland (Unknown); University of Lausanne Hospitals (Other); Department of Neonatology, University Hospital Geneva (HUG), Switzerland (Unknown); Division of Development and Growth, University Hospital Geneva (HUG), Switzerland (Unknown); Neonatal and Paediatric Intensive Care Unit, Children's Hospital of Lucerne, Switzerland (Unknown); Department of Pediatrics, Cantonal Hospital Muensterlingen, Switzerland (Unknown); Department of Pediatrics, Cantonal Hospital Neuchatel, Switzerland (Unknown); Cantonal Hospital of St. Gallen (Other); Department of Child Development, Children's Hospital St. Gallen, Switzerland (Unknown); Department of Neonatology, Cantonal Hospital Winterthur, Switzerland (Unknown); Social Pediatrics Center, Cantonal Hospital Winterthur, Switzerland (Unknown); University Hospital, Zürich (Other); University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2016-02299
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Very Low Birth Weight Infant; Very Preterm Maturity of Infant; Asphyxia Neonatorum
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Minimal Neonatal Dataset MNDS: All Swiss live-born infants below 32 weeks gestational age or 1501g birth weight
- Below 34, B34: All Swiss live-born infants between 32 0/1 and 33 6/7 weeks gestational age that are above 1500g birth weight
- Swiss Asphyxia and Cooling Registry, ASP: Infants between 35 0/7 and 42 6/7 weeks' gestational age with moderate or severe encephalopathy due to perinatal asphyxia

SUMMARY:
The chief aim of the Swiss Neonatal Network & Follow-Up Group (SwissNeoNet) is to maintain and / or improve the quality and safety of medical care for high-risk newborn infants and their families in Switzerland through a coordinated program of research, education and collaborative audit. In support of its aim, SwissNeoNet hosts the official medical quality register for the Swiss level III and level IIB units. Participation for these units is mandatory according to the intercantonal declaration for Highly Specialized Medicine (HSM) of September 22, 2011 and the Society's Standards for Levels of Neonatal Care in Switzerland.

DETAILED DESCRIPTION:
Inaugurated in 1995, SwissNeoNet now routinely collects data from 9 level III, 10 level IIB and 14 neuro-/developmental pediatric units encompassing information about the care and outcomes of high-risk newborn infants. Data collection is monitored for population coverage, dataset completeness, plausibility and reliability. Data quality is audited within a three year cycle.

Quality improvement

SwissNeoNet releases an annual quality report for participating centers encompassing up to 20 process- and outcome quality indicators. It annually collects data on unit infrastructure evaluated by the Committee for the Accreditation of Neonatology Units (CANU). To discuss quality issues and educational purposes, it hosts bi-annual meetings/symposia for the NEO Directors Group and the Follow-up Group, respectively. The SwissNeoNet member platform offers tools for unit-to-unit quality improvement collaboration (mailing lists, event-organizer, forum, file-sharing and survey builder).

Research

SwissNeoNet coordinates cross-sectional and longitudinal cohort studies that are performed by local researchers using SwissNeoNet's prospectively collected data. These studies focus on mortality, morbidity and/or long-term outcome issues and the analysis of risk factors for development. The network disseminates its research in scientific articles in peer reviewed medical journals.

Support

SwissNeoNet supports the units logistically to ensure that each patient receives primary care (NICU bed availability) and follow-up assessments at 9 to 12 months corrected, 18 to 24 months corrected, and at 5.5 to 6 years of age (FU missing lists) to ensure early diagnosis and intervention. With regards to its Follow-up program, the SwissNeoNet also supports training of new staff and coordinates the launch of new testing instruments between centers.

ELIGIBILITY:
Inclusion criteria of "Minimal Neonatal Dataset" (MNDS):

All Swiss live-born infants below 32 weeks gestational age or 1501g birth weight

Inclusion criteria of "Below 34 data collection", (B34):

All Swiss live-born infants between 32 0/1 and 33 6/7 weeks gestational age that are above 1500g birth weight

Inclusion criteria of "Swiss Asphyxia and Cooling Registry", (ASP):

Infants between 35 0/7 and 42 6/7 weeks' gestational age with moderate or severe encephalopathy due to perinatal asphyxia

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: see cohort descriptions under 'Groups and Interventions'
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 0 to 6 years
  Mortality in delivery room, during primary hospitalization or within first 6 years of life
Major morbidities of newborns | 0 to 6 years
  Period prevalences (i.e. incident proportions per year or period of years) of intraventricular hemorrhages, necrotizing enterocolitis, sepsis, retinopathy of prematurity, bronchopulmonary displasia, neurodevelopmental impairment at 2 or 6 years, and other

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SwissNeoNet description — https://www.neonet.ch/swissneonet/aims-and-description
- See also: SwissNeoNet publications — https://www.neonet.ch/swissneonet/publications